CLINICAL TRIAL: NCT03556254
Title: Comparison of Genotypic Resistance Guided Versus Susceptibility Testing Guided Therapy for the First-line Eradication of H. Pylori- a Multicenter Randomized Trial
Brief Title: Genotypic Resistance Guided Versus Susceptibility Testing Guided Therapy for the First-line Eradication of H. Pylori
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201706038MINC
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; Genotypic resistance; Antimicrobial susceptibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotypic resistance guided therapy (Experimental): In the absence of 23S rRNA mutation, clarithromycin based sequential therapy will be given. In the presence of 23S rRAN mutation but the absence of gyrase A mutation, levofloxacin based sequential therapy will be given. In the presence of both 23S rRNA and gyrase A mutations or if genotyping fails, bismuth quadruple therapy will be given.
  Interventions: Drug: GGT
- Susceptibility testing guided therapy (Active Comparator): Tailored therapy according to the minimum inhibitory concentration result (susceptibility testing, E-test)
  Interventions: Drug: SGT

INTERVENTIONS:
Drug: GGT — In the absence of 23S rRNA mutation, clarithromycin based sequential therapy will be given. In the presence of 23S rRAN mutation but the absence of gyrase A mutation, levofloxacin based sequential therapy will be given. In the presence of both 23S rRNA and gyrase A mutations or if genotyping fails, bismuth quadruple therapy will be given
  Arms: Genotypic resistance guided therapy
Drug: SGT — In the absence of clarithromycin resistance, clarithromycin based sequential therapy will be given. In the presence of clarithromycin resistance but the absence of levofloxacin resistance, levofloxacin based sequential therapy will be given. In the presence of both clarithromycin and levofloxacin resistance or if culture fails, bismuth quadruple therapy will be given.
  Arms: Susceptibility testing guided therapy

SUMMARY:
We aimed to (1) compare the efficacy of genotypic resistance guided sequential therapy vs. susceptibility testing guided therapy in the first-line therapy (2) assess the long term impact of eradication therapy on the antibiotic resistance and microbiota of the gut flora and the metabolic factors in this multi-center, open labeled trial

DETAILED DESCRIPTION:
Background: Recent trials have shown that susceptibility testing guided therapy was more effective than empirical triple therapy given for 7-10 days in the first-line treatment of H. pylori infection. However, susceptibility testing is time consuming and inconvenient, limiting the widespread application of susceptibility testing guided therapy in clinical practice. Recently, point mutations at 23S rRNA and gyrase A have reported to be associated with clarithromycin and levofloxacin resistance. However, whether genotypic resistance guided therapy is more effective or non-inferior to susceptibility guided therapy has not been reported. Besides, the long term impact of H. pylori eradication on the gut microbiota and metabolic disorders remains unclear. Aim: Therefore, we aimed to (1) compare the efficacy of genotypic resistance guided sequential therapy vs. susceptibility testing guided therapy in the first-line therapy(2) assess the long term impact of eradication therapy on the antibiotic resistance and microbiota of the gut flora and the metabolic factorsMethods: This will be a multi-center, open labeled trialPatients: 560 patients with H. pylori infection naïve to eradication therapy will be enrolled Testing for H. pylori infectionBefore First Line TreatmentAny two positive of CLO test, histology, HpSA, and culture will be considered as H. pylori infectedAfter First-Line Treatment: C13-UBT will be used to assess the existence of H. pylori 6-8 weeks after first line therapy. Long term reinfection: C13-UBT will be used to assess the recurrence of H. pylori 1 year after eradication therapy Determination of antibiotic resistance of H. pylori: E-test will be used to determine the minimum inhibitory concentrations of clarithromycin and levofloxacin to guide the selection of antibiotics. Agar dilution test will also be done. Mutations in 23S rRNA and gyrase A will also be determined by PCR followed by direct sequencing Treatment regimens and assignment Eligible patients will be randomized to receive either one of the treatments (A) Genotypic resistance guided therapy: In the absence of 23S rRNA mutation, clarithromycin based sequential therapy will be given. In the presence of 23S rRAN mutation but the absence of gyrase A mutation, levofloxacin based sequential therapy will be given. In the presence of both 23S rRNA and gyrase A mutations or if genotyping fails, bismuth quadruple therapy will be given. (B) Susceptibility testing guided therapy: In the absence of clarithromycin resistance, clarithromycin based sequential therapy will be given. In the presence of clarithromycin resistance but the absence of levofloxacin resistance, levofloxacin based sequential therapy will be given. In the presence of both clarithromycin and levofloxacin resistance or if culture fails, bismuth quadruple therapy will be given. The stool samples will be collected before, and 2 and 8 weeks and 1 year after eradication therapy to analyze the changes in the antibiotic resistance and microbiota of gut floraThe body weight, waist and hip circumference and serum lipid profile, sugar, and HbA1C levels will be collected before and 8 weeks and 1 year after eradication therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged greater than 20 years with H. pylori infection naïve to treatment are considered eligible for enrollment..

Exclusion Criteria:

* children and teenagers aged less than 20 years
* history of gastrectomy
* gastric malignancy, including adenocarcinoma and lymphoma
* previous allergic reaction to antibiotics (amoxicillin, clarithromycin, levofloxacin, metronidazole, bismuth) and prompt pump inhibitors (esomeprazole)
* contraindication to treatment drugs
* pregnant or lactating women
* severe concurrent disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate will be evaluated according to Intent-to-treat (ITT) analyses | 6 weeks
  Urea breath testing will be done at least 6 weeks after completion of eradication therapy

SECONDARY OUTCOMES:
adverse effects during eradication therapies | 2 weeks
  a standard interview will be arranged at the end of treatment to assess the adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Yun-Lin County, Taiwan

REFERENCES:
- [Derived] Chen MJ, Chen PY, Fang YJ, Bair MJ, Chen CC, Chen CC, Yang TH, Lee JY, Yu CC, Kuo CC, Chiu MC, Chou CK, Chen CY, Hu WH, Tsai MH, Hsu YC, Shun CT, Luo JC, Lin JT, El-Omar EM, Wu MS, Liou JM; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Molecular testing-guided therapy versus susceptibility testing-guided therapy in first-line and third-line Helicobacter pylori eradication: two multicentre, open-label, randomised controlled, non-inferiority trials. Lancet Gastroenterol Hepatol. 2023 Jul;8(7):623-634. doi: 10.1016/S2468-1253(23)00097-3. Epub 2023 May 10. PMID 37178702